CLINICAL TRIAL: NCT07385170
Title: Evaluation of Perioperative Continuous Glucose Monitoring Accuracy in Patients Undergoing Cardiac Surgery
Brief Title: Perioperative Continuous Glucose Monitoring Accuracy in Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Karam Nam, MD, Clinical Associate Professor, Seoul National University Hospital
Other Study IDs: CGM-CS
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery
Keywords: continuous glucose monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CGM cohort: Application of perioperative continuous glucose monitoring
  Interventions: Device: Dexcom G7

INTERVENTIONS:
Device: Dexcom G7 — Continuous glucose monitoring device (Dexcom G7) will be applied to patients undergoing cardiac surgery intraoperatively and postoperatively (maximum 10 days)

SUMMARY:
The goal of this clinical trial is to evaluate accuracy of continuous glucose monitoring device called 'Dexcom G7' in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older scheduled for cardiac surgery

Exclusion Criteria:

* Skin disease at the sensor application site (proximal arm)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who scheduled for cardiac surgery in Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
MARD | From the beginning of operation to the end of postoperative ICU stay (maximum 10 days)
  mean absolute relative difference

SECONDARY OUTCOMES:
Bland-Altman analysis | From the beginning of operation to the end of postoperative ICU stay (maximum 10 days)
  mean difference, bias, 95% limits of agreement
ISO criteria | From the beginning of operation to the end of postoperative ICU stay (maximum 10 days)
  Satisfaction of 2013 ISO (International Organization of Standardization) criteria
DTS error grid | From the beginning of operation to the end of postoperative ICU stay (maximum 10 days)
  DTS (Diabtetes Technology Society) error grid

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No